CLINICAL TRIAL: NCT02442219
Title: A Blood Based Diagnostic Test for Coeliac Disease
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Associate professor, phD, MD, Oslo University Hospital
Other Study IDs: 2011/2472
Record Dates: First submitted 2015-04-15; First posted 2015-05-13 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Coeliac Disease; Non Coeliac Gluten Sensitivity
Keywords: gluten; Tetramer
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A tetramerbased bloodtest which will bind and identify gluten specific T-cells by the use of a flow cytometer. 50 ml blood will be needed for this test, along with characterization of other blood values (eg. Hb, leukocytes, transferrin binding, B12, biobanking etc).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Coeliac: Persons with coeliac disease on a gluten free diet where diagnosis is confirmed by duodenal biopsy.
- Non coeliac gluten sensitive: Persons on a gluten free diet where coeliac disease is excluded by duodenal biopsy.
- Healthy control group: Persons on a gluten containing diet without known coeliac disease.

SUMMARY:
Persons with coeliac disease treated with a gluten free diet will be asked to give blood for a new diagnostic blood test. In this test investigators will use multimerized HLA bound to different gliadin-peptides (tetramer) and with the help of a flow-cytometer identify (along with other relevant T-cell-markers) gluten specific T-cells. Investigators believe that these cells will be present in persons with coeliac disease regardless of gluten-intake. Investigators will compare their findings with two control groups; Persons on a gluten free diet where celiac disease is excluded (gluten sensitive group) and persons on a gluten containing diet (healthy control group). In the initial and main study investigators will look at HLA DQ2.5 individuals, which comprise >90% of all persons with coeliac disease.

ELIGIBILITY:
Inclusion Criteria:

* HLA DQ2.5 positives in primary blinded study (other HLA-types ie DQ8 and DQ2.2 in later unblinded study)
* In gluten free group: Diagnosis must be confirmed by duodenal biopsy done after sufficient time on gluten containing diet and participant must have followed a glutenfree diet since.

Exclusion Criteria:

* Drugs that influence the immune system used last three months
* Infected with Hepatitis B, C or HIV
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are invited through announcement in media. Eligibility is tested through HLA-test and previous workup with confirmation / exclusion of coeliac disease by reference method (duodenal biopsy).
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Ability of the tetramer test in differentiating persons with coeliac disease from controls by the use of tetramer staining for gluten specific T-cells and flowcytometry | Upto 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Knut EA Ludin, PhD, MD, Principal Investigator — University of Oslo. Oslo University Hospital.
Locations (1):
- Oslo University hospital, Oslo, Norway

REFERENCES:
- [Derived] Sarna VK, Lundin KEA, Morkrid L, Qiao SW, Sollid LM, Christophersen A. HLA-DQ-Gluten Tetramer Blood Test Accurately Identifies Patients With and Without Celiac Disease in Absence of Gluten Consumption. Gastroenterology. 2018 Mar;154(4):886-896.e6. doi: 10.1053/j.gastro.2017.11.006. Epub 2017 Nov 14. PMID 29146521